CLINICAL TRIAL: NCT04868760
Title: Compare IBI310 and Ipilimumab on the Pharmacokinetics, Safety, Tolerance and Immunogenicity of a Single Dose In Healthy Male Subjects: a Randomized Double-blind Parallel Controlled Phase I Clinical Study
Brief Title: A Study to Evaluate the Similarity in Pharmacokinetics and Safety of IBI310 and Ipilimumab（YERVOY）in Adult Healthy Chinese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIBI310G101
Record Dates: First submitted 2021-04-23; First posted 2021-05-03 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2022-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Ipilimumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B: ipilimumab (Active Comparator): Ipilimumab, 0.1 and 0.3mg/kg, will be administrated intravenously in 30-60 minutes.
  Interventions: Drug: Ipilimumab
- Group A: IBI310 (Experimental): IBI 310, 0.1 and 0.3mg/kg, will be administrated intravenously in 30-60 minutes.
  Interventions: Drug: IBI310

INTERVENTIONS:
Drug: Ipilimumab — Drug: Ipilimumab 0.1 mg/kg and 0.3 mg/kg in preparatory experiments and 0.3 mg/kg in formal experiment.
  Arms: Group B: ipilimumab
Drug: IBI310 — Drug: IBI310 0.1 mg/kg and 0.3 mg/kg in preparatory experiments and 0.3 mg/kg in formal experiment.
  Arms: Group A: IBI310

SUMMARY:
This trail will investigate the pharmacokinetics and safety of IBI310 and establish pharmacokinetics biosimilarity of IBI310 to ipilimumab （YERVOY）

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, patients should fulfill all the following criteria:

1. Fully understand the study purpose, and understand the pharmacological effects and potential adverse reactions of the drug, voluntarily signed written informed consent according to the declaration of Helsinki.
2. Aged 18-55 years healthy male subjects
3. Weigh ranges from 50-80 kg， BMI ranges from 19.0-28.0 kg/m2
4. All the system test result within the normal range, or abnormal test results without clinical significance judged by the investigator.
5. The subjects must agree to use effective contraceptive measures during the study treatment and for 6 months after receiving last does of study drug (e.g. abstinence, sterilization surgery, oral contraceptives, contraception by progesterone injection or subcutaneous)

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Medical history of chronic liver, kidney, cardiovascular, neurological/psychiatric, digestive tract, respiratory, urinary, endocrine and other system diseases;
2. Medical history of autoimmune diseases (see Annex 1);
3. People who drink frequently in the 6 months before screening (the definition of frequent drinking is defined as drinking more than 2 units per day on average, or drinking more than 14 units of alcohol per week on average: 1 unit = 360ml of beer or 45ml of alcohol is 40 % Of spirits or 150ml wine);
4. Have opportunistic infections within 6 months before screening (such as: herpes zoster, active cytomegalovirus, pneumocystis carinii, histoplasma, aspergillus, mycobacterium, etc.)
5. Medical history of recurrence or chronic infection, have had chronic or recurrent infections, including but not limited to: chronic kidney infection, chronic chest infection (such as bronchiectasis), sinusitis, recurrent urinary tract infections, those with open, draining or infected skin wounds;
6. Acute infection within 2 weeks before screening;
7. Medical history of malignant tumors, unless they are squamous cell carcinoma of the skin, basal cell carcinoma or local cervical carcinoma in situ that have been successfully removed and have no evidence of metastasis;
8. Suspected or confirmed to be allergic or have experienced severe drug or food allergic reactions in the past, have clear history of allergies and/or are allergic to test drugs or their ingredients;
9. Any drugs (including Chinese medicines and vitamins) have been used within 2 weeks before the screening, or the last dose is less than 5 half-lives of the drug from the trial dosing day, whichever is longe;
10. Any prior using of ipilimumab;
11. Participation in any other interventional clinical trials within 3 months before screening;
12. Subjects have made a blood donation or a comparable blood lossor received any blood transfusion (>400 mL) within the last 3 months prior to screening.
13. Subjects underwent major surgery or hospitalization for illness within 3 months before screening;
14. Subjects have received live vaccines within 6 months prior to screening, or expect to receive live vaccines during the study period;
15. Any drug abuse or positive drug screening result within 12 months before screening;
16. Any abnormalities of vital signs and physical examination with clinical significance as judged by investigators at screening;
17. Abnormalities in the ECG with clinicavl significance judged by investigators at screening;
18. Abnormalities of chest-X ray or CT examination with clinical significance as judged by investigators at screening;
19. Abnormal laboratory tests with clinical significance at screening.
20. Known Tuberculosis (TB) disease, high risk of acquiring TB infection, or latent TB infection (including but not limited to tuberculosis, lymphatic tuberculosis, tuberculous pleurisy, etc.), tuberculosis laboratory examination (QuantiFERON-TB tuberculosis test/T.SPOT tuberculosis test) is positive.
21. Human Immunodeficiency Virus (HIV) antibody, Hepatitis C virus (HCV) antibody, Syphilis test (RPR), Hepatitis B virus (HBV) surface antigen, e antigen ( HBeAg) or core antibody (HBcAb) is positive;
22. Have a childbirth plan within 6 months from the screening period to the trial drug administration, or who are unwilling to take the contraceptive measures specified in the protocol during the trial period;
23. It is not suitable to participate in this clinical trial due to other reasons per investigator discretion

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve (AUC0-inf) | From pre-dose to 1848hrs (78day)
Maximum Plasma Concentration (Cmax) | From pre-dose to 1848hrs (78day)

SECONDARY OUTCOMES:
Area Under the Concentration-time Curve | From pre-dose to 1848hrs (78day)
Clearance | From pre-dose to 1848hrs (78day)
Volume of distribution | From pre-dose to 1848hrs (78day)
Positive rate of ADA and Nab | From pre-dose to 1848hrs (78day)
incidence and severity of adverse events | from dosing to completion of study (183days posy-dosing) or to the patient withdrawl
  Number of subjects with AE，treatment-related AE (TRAE), immune-related AEs (irAE), serious adverse SAE assessed by CTCAE V5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, China